CLINICAL TRIAL: NCT04395612
Title: A Clinical Proof-of-concept Study Evaluating Efficacy and Safety of ZL-2306 (Niraparib) Combined With Brivanib or Toripalimab in Patients With Metastatic, Recurrent, and Persistent Cervical Cancer
Brief Title: Niraparib Combined With Brivanib or Toripalimab in Patients With Cervical Cancer
Acronym: CQGOG0101
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chongqing University Cancer Hospital (Other)
Responsible Party: Principal Investigator, Qi Zhou, Professor, Chongqing University Cancer Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CQGOG0101
Record Dates: First submitted 2020-04-23; First posted 2020-05-20 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-03

CONDITIONS: Cervical Cancer
Keywords: Cervical Cancer,Niraparib,Brivanib,Toripalimab
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — brivanib; toripalimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment arm1 (Experimental): niraparib 200mg/day and brivanib 400mg/day
  Interventions: Drug: niraparib combined with brivanib
- Treatment arm2 (Experimental): niraparib 200mg/day and toripalimab 240mg/21 days
  Interventions: Drug: niraparib combined with toripalimab

INTERVENTIONS:
Drug: niraparib combined with brivanib — Drug：Niraparib will be administered as a dose of 200 mg orally every day. Drug：Brivanib will be administered as a dose of 400mg orally every day.
  Other Names: Treatment group1
  Arms: Treatment arm1
Drug: niraparib combined with toripalimab — Drug：Niraparib will be administered as a dose of 200 mg orally every day. Drug：Toripalimab will be administered as a dose of 240mg Intravenously every 21days.
  Other Names: Treatment group2
  Arms: Treatment arm2

SUMMARY:
A Clinical Proof-of-concept Study Evaluating Efficacy and Safety of ZL-2306 (Niraparib) Combined With Brivanib or Toripalimab in Patients With Metastatic, Recurrent, and Persistent Cervical Cancer

DETAILED DESCRIPTION:
A prospective, open-ended, single-arm, phase II clinical study.Patients are with metastatic, recurrent, persistent cervical cancer (squamous cell carcinoma, adenocarcinoma, adenosquamous carcinoma) To observe the efficacy and safety of ZL-2306 (Niraparib) combined with Brivanib or Toripalimab in patients with metastatic, recurrent and persistent cervical cancer, and to explore the biomarkers of effectiveness.

ELIGIBILITY:
Inclusion Criteria:

1. Female, aged ≥ 18 yrs and ≤70 yrs;
2. Patients volunteered to participate in this study, signed informed consent, good compliance, and cooperated with follow-up;
3. The subjects' damage caused by other treatments has been recovered (NCI CTCAE version 5.0 grade ≤ grade 1), ECOG score ≤ 2 points
4. Expected survival is longer than 3 months;
5. Pathological diagnosis of cervical squamous cell carcinoma, adenocarcinoma, and adenosquamous carcinoma;
6. Evaluable lesions: CT scan of tumor lesions ≥5mm in length, CT scan of lymph node lesions ≥10mm in length, and scan layer thickness not greater than 5mm (refer to RECIST 1.1);
7. The first diagnosis was confirmed by pathology and / or cytology to be metastatic, or recurrent, persistent cervical cancer (mainly refers to tumors remaining or progressing at least 3 months after initial radiotherapy or concurrent chemoradiotherapy), and the patient can no longer accept Surgery or chemoradiation;
8. Subject agrees to take blood sample;
9. Subjects can provide formalin-fixed, paraffin-embedded tumor tissue samples for subsequent related gene testing (optional);
10. A.Complete blood count: hemoglobin (Hb) ≥90g/L ; absolute neutrophil count (ANC) ≥1.0×109/L ; platelets >=100×109/L B. Biochemical test standards: a. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2 times the upper limit of normal value (ULN). If with liver metastases, ALT and AST ≤ 5 × ULN; b. Total bilirubin (TBIL) ≤ 1.5 × ULN; c. Serum creatinine (Cr) ≤ 1.5 × ULN or creatinine clearance (CCr) ≥ 60ml / min; d. Doppler ultrasound evaluation: left ventricular ejection Blood fraction (LVEF) ≥ the lower limit of normal value (50%).
11. Women of childbearing age should agree that contraception (such as an intrauterine device, contraceptive, or condom) must be used during the study and within 3 months after the last dose; a serum or urine pregnancy test must be negative within 14 days of study enrollment and must be Non-lactating patients. Sign written informed consent before conducting any research-related procedures.

Exclusion Criteria:

* 1.People who are known to be allergic to zl-2306 (niraparib)，brivanib and toripalimab or to active or inactive ingredients of drugs with similar chemical structures to zl-2306 (niraparib），brivanib and toripalimab.

  2.Multiple factors affecting oral medication (such as inability to swallow, post-gastrointestinal resection, chronic diarrhea, etc.).

  3.Symptomatic, uncontrolled brain metastases or pia meningeal metastases. No imaging scan is required to confirm brain-free metastases; patients with spinal cord compression may still be considered if they have received targeted treatment and have evidence of clinical stability of the disease for at least> 28 days (controlled central nervous system metastasis must be in the study Have received treatment such as radiation or chemotherapy for at least 1 month; patients must not have new symptoms related to central nervous system lesions or symptoms that indicate disease progression, and patients either take a stable dose of hormones or do not need to take hormones).

  5.Underwent major surgery within 3 weeks before the study began, or any surgical effects that have not recovered after surgery, or received chemotherapy.

  6.Received> 20% bone marrow palliative radiotherapy 1 week before enrollment. 7.Have aggressive cancers other than cervical cancer (except fully treated basal or squamous cell skin cancer within 2 years before enrollment).

  8.Patient has a previous or current diagnosis of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML).

  9.Suffering from a serious or uncontrolled illness, including but not limited to:
  1. Uncontrollable nausea and vomiting, inability to swallow research drugs, and any gastrointestinal disorders that may interfere with the metabolism of the drug.
  2. Active viral infections such as human immunodeficiency virus, hepatitis B, hepatitis C, etc.
  3. Uncontrolled major seizures, unstable spinal cord compression, superior vena cava syndrome, or other mental illnesses that prevent patients from signing informed consent.
  4. Immunodeficiency (except splenectomy), or other diseases that the investigator believes may expose patients to high-risk toxicity.

     10.History of bleeding and thrombosis:

  <!-- -->

  1. Any CTCAE Grade 2 bleeding event within 3 months prior to screening, or CTCAE Grade 3 and above bleeding events within 6 months prior to screening.
  2. History of gastrointestinal bleeding or clear gastrointestinal bleeding tendency within 6 months before screening. Such as: esophageal varices at risk of bleeding, focal lesions of locally active ulcers, or fecal occult blood +.
  3. Have active bleeding or coagulopathy, have a tendency to bleed, or are receiving thrombolytic or anticoagulant therapy.
  4. Patients need anticoagulation with drugs such as warfarin or heparin.
  5. Patients need long-term antiplatelet therapy (eg aspirin, clopidogrel).
  6. Thrombosis or embolism events in the past 6 months, such as: cerebrovascular accidents (including transient ischemic attacks), pulmonary embolism.

     11.Serious cardiovascular history:

  <!-- -->

  1. NYHA (New York Heart Association) Grade 3 and 4 congestive heart failure.
  2. Suffering from unstable angina or newly diagnosed angina or myocardial infarction within 12 months before screening.
  3. Arrhythmias requiring therapeutic intervention (patients taking beta-blockers or digoxin can be enrolled).
  4. CTCAE≥ grade 2 valvular heart disease.

     12.Poorly controlled hypertension (systolic blood pressure> 150 mmHg or diastolic blood pressure> 100 mmHg).

     13.Other laboratory inspection abnormalities:

  <!-- -->

  1. Hyponatremia (sodium <130 mmol / L); baseline serum potassium <3.5 mmol / L (before entering the study, potassium supplements can be used to restore serum potassium above this level).
  2. Abnormal thyroid function, and drugs cannot maintain thyroid function within normal range.

     14.Any previous or current disease, treatment, or laboratory abnormality that may interfere with the results of the study, affect the patient's full participation in the study, or the investigator believes that the patient is not suitable to participate in the study; the patient may not receive platelets within 4 weeks before the study drug begins Red blood cell infusion.

     15.Patients who are pregnant or breastfeeding, or plan to become pregnant during study treatment.

     16.Corrected QTc interval (QTc)> 450 milliseconds; if the patient has a prolonged QTc interval, but the investigator evaluates that the reason for the prolongation is a pacemaker (and no other cardiac abnormalities), it is necessary to discuss with the investigator to determine whether the patient is suitable Group study.

     17.With any active autoimmune disease or have a history of autoimmune disease (including but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism, hypothyroidism; patients with vitiligo or asthma has been completely relieved in childhood and do not need any intervention after adulthood could be included; Asthma patient who need bronchodilators for medical intervention cannot be included) 18.Treatment with other immunosuppressive medications, systemic or topical corticosteroids (>10 mg daily prednisone or equivalent) within 14 days before enrollment.

     19.With a history of severe allergic reaction to other monoclonal antibodies 20.Evidence of central nervous system metastasis (such as brain edema requiring hormone intervention, or brain metastasis progression). Patients who have previously received treatment for brain or meningeal metastasis and persistently stable (MRI) for at least 1 month thus stopped systemic hormone therapy (dose > 10mg/ prednisone or other therapeutic hormones) for more than 2 weeks can be included.

     21.Have previously received any PARP inhibitor or PD-1/PD-L1 inhibitor treatment.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2020-05-08 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
ORR | 6 months
  Objective To evaluate the objective response rate (CR + PR) of ZL-2306 (niraparib) combined with brivanib or toripalimab in patients with relapsed and persistent cervical cancer.

SECONDARY OUTCOMES:
PFS | 6 months
  progression-free survival
DCR | 6 months
  evaluate the safety of combined application of ZL-2306 (niraparib) combined with brivanib or toripalimab， disease control rate

CONTACTS AND LOCATIONS:
Overall Officials: Qi Zhou, Ph.D., Principal Investigator — Chongqing University Cancer Hospital
Locations (1):
- Chongqing Cancer Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mirza MR, Monk BJ, Herrstedt J, Oza AM, Mahner S, Redondo A, Fabbro M, Ledermann JA, Lorusso D, Vergote I, Ben-Baruch NE, Marth C, Madry R, Christensen RD, Berek JS, Dorum A, Tinker AV, du Bois A, Gonzalez-Martin A, Follana P, Benigno B, Rosenberg P, Gilbert L, Rimel BJ, Buscema J, Balser JP, Agarwal S, Matulonis UA; ENGOT-OV16/NOVA Investigators. Niraparib Maintenance Therapy in Platinum-Sensitive, Recurrent Ovarian Cancer. N Engl J Med. 2016 Dec 1;375(22):2154-2164. doi: 10.1056/NEJMoa1611310. Epub 2016 Oct 7. PMID 27717299
- [Result] Torre LA, Bray F, Siegel RL, Ferlay J, Lortet-Tieulent J, Jemal A. Global cancer statistics, 2012. CA Cancer J Clin. 2015 Mar;65(2):87-108. doi: 10.3322/caac.21262. Epub 2015 Feb 4. PMID 25651787
- [Result] Chen WQ, Li H, Sun KX, Zheng RS, Zhang SW, Zeng HM, Zou XN, Gu XY, He J. [Report of Cancer Incidence and Mortality in China, 2014]. Zhonghua Zhong Liu Za Zhi. 2018 Jan 23;40(1):5-13. doi: 10.3760/cma.j.issn.0253-3766.2018.01.002. Chinese. PMID 29365411
- [Result] Eskander RN, Tewari KS. Immunotherapy: an evolving paradigm in the treatment of advanced cervical cancer. Clin Ther. 2015 Jan 1;37(1):20-38. doi: 10.1016/j.clinthera.2014.11.010. PMID 25592089
- [Result] Kaelin WG Jr. The concept of synthetic lethality in the context of anticancer therapy. Nat Rev Cancer. 2005 Sep;5(9):689-98. doi: 10.1038/nrc1691. PMID 16110319
- [Result] Chu JS, Ge FJ, Zhang B, Wang Y, Silvestris N, Liu LJ, Zhao CH, Lin L, Brunetti AE, Fu YL, Wang J, Paradiso A, Xu JM. Expression and prognostic value of VEGFR-2, PDGFR-beta, and c-Met in advanced hepatocellular carcinoma. J Exp Clin Cancer Res. 2013 Apr 3;32(1):16. doi: 10.1186/1756-9966-32-16. PMID 23552472
- [Result] Kirstein MM, Lange A, Prenzler A, Manns MP, Kubicka S, Vogel A. Targeted therapies in metastatic colorectal cancer: a systematic review and assessment of currently available data. Oncologist. 2014 Nov;19(11):1156-68. doi: 10.1634/theoncologist.2014-0032. Epub 2014 Oct 17. PMID 25326159
- [Result] Fakhrejahani E, Toi M. Antiangiogenesis therapy for breast cancer: an update and perspectives from clinical trials. Jpn J Clin Oncol. 2014 Mar;44(3):197-207. doi: 10.1093/jjco/hyt201. Epub 2014 Jan 27. PMID 24474817